CLINICAL TRIAL: NCT00439946
Title: Rapid Switch From Intravenous Epoprostenol to Intravenous Remodulin® (Treprostinil Sodium) Using the Crono Five Ambulatory Infusion Pump in Patients With Stable Pulmonary Arterial Hypertension (PAH): Safety, Efficacy and Treatment Satisfaction
Brief Title: Safety, Efficacy, and Treatment Satisfaction Switching From Flolan to Remodulin Using the Crono Five Ambulatory Pump in Patients With PAH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study closed due to limited availability of eligible subjects and competition by for enrollment by other studies
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIV-PH-410
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Results first posted 2013-07-17 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2013-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary hypertension; PAH; Remodulin; treprostinil; Quality of Life; rapid switch
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treprostinil (Experimental): IV treprostinil continuous infusion via Crono Five infusion pump.
  Interventions: Drug: treprostinil; Device: Crono Five ambulatory pump

INTERVENTIONS:
Drug: treprostinil — rapid switch from intravenous epoprostenol on the CADD ambulatory pump to intravenous Remodulin on the Crono Five ambulatory pump
  Other Names: Remodulin
Device: Crono Five ambulatory pump — Used for administration of IV Remodulin (treprostinil)

SUMMARY:
The purpose of this 8-week study is to compare the effects of switching from intravenous Flolan to intravenous Remodulin therapy. Remodulin (treprostinil sodium) is an approved therapy for pulmonary arterial hypertension (PAH). Unlike Flolan, Remodulin does not need to be mixed daily and is stable at room temperature, so there is no need for ice packs. In addition, Remodulin is changed every 48hrs, instead of every 12-24 (with ice packs) or every 8 hours (without ice packs) with Flolan. Flolan is given using a type of portable medication pump called the CADD Legacy infusion pump. In this study, Remodulin will be given using a smaller and lighter medication pump called the Crono Five infusion pump. This study will also assess the effect that changing to Remodulin will have on treatment satisfaction and patient quality of life.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH), which is defined as an elevation in pulmonary arterial pressure and pulmonary vascular resistance, is a severe hemodynamic abnormality common to a variety of diseases and syndromes. Elevation in pulmonary arterial pressure causes an increase in right ventricular afterload, impairing right ventricular function and ultimately leading to inactivity and death. The goal of PAH treatment is to lengthen survival time, to ameliorate symptoms of PAH, and to improve health related quality of life (HRQOL).

Remodulin® (treprostinil sodium), a stable analogue of prostacyclin, possesses potent pulmonary and systemic vasodilatory and platelet anti-aggregatory actions in vitro and in vivo. Recently, Remodulin received FDA approval for intravenous therapy based upon bioequivalence of the intravenous (IV) and subcutaneous (SC) routes of administration. Remodulin is more chemically stable than epoprostenol and may offer potential safety and convenience advantages compared to intravenous epoprostenol that may impact Health Related Quality of Life (HRQOL) and/or patient satisfaction. Unlike epoprostenol, Remodulin does not need to be mixed daily and is stable at room temperature eliminating the need for ice packs. Since Remodulin remains in the body longer than epoprostenol (4 hrs instead of less than 5 minutes) there is less risk of cardiovascular collapse from a sudden interruption of infusion, such as a line clog. In an open-label study in Europe, patients who were using a type of portable medication pump called the CADD Legacy pump were rapidly switched from Flolan to Remodulin with no serious side effects. This study will examine effects of switching from therapy with epoprostenol or Flolan to IV Remodulin and compare changes in HRQOL and treatment satisfaction before and after rapid switch from epoprostenol to Remodulin in patients with pulmonary hypertension from the CADD legacy pump to a smaller pump called the Crono Five.

Participation in this study will last approximately 10 weeks. Study procedures include routine blood tests, medical history, physical exams, disease evaluation, exercise tests and patient questionnaires. Participants will have 4 visits during the study and will spend at least 1 night in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Diagnosis of one of the following WHO Classifications of pulmonary hypertension:

  1. Group 1 pulmonary arterial hypertension

     * Idiopathic pulmonary arterial hypertension (IPAH)
     * Familial pulmonary arterial hypertension (FPAH)
     * Associated pulmonary arterial hypertension (APAH):

       1. collagen vascular disease
       2. congenital systemic-to-pulmonary shunt repaired greater than 5 years prior to study entry.
       3. portal hypertension
       4. drugs and toxins
  2. Group 4 pulmonary hypertension due to chronic thromboembolic pulmonary hypertension (CTEPH)
* WHO Class II-III
* Currently receiving intravenous epoprostenol therapy for at least three months and a stable dose for at least one month.
* Have central intravenous catheter
* Optimally treated with conventional pulmonary hypertension therapy and clinically stable for at least one month.
* Mentally and physically capable of learning to administer Remodulin using an intravenous infusion pump.

Exclusion Criteria:

* nursing or pregnant woman
* received a new type of chronic therapy (including but not limited to oxygen, a different category of vasodilator, a diuretic, digoxin, bosentan, sildenafil) for pulmonary hypertension added within the last month.
* Had any PAH medication discontinued within the week prior to study entry.
* Received any prostacyclin or prostacyclin analog except epoprostenol in the past 3 months.
* Had a central venous line infection within the past 30 days.
* Previous documented evidence of significant parenchymal lung disease as evidenced by pulmonary function tests as follows (any one of the following):

  1. Total Lung Capacity ≤ 60% (predicted) or
  2. If Total Lung Capacity is between 60% and 70% (predicted), a High Resolution Computed Tomography (CT) scan must be performed to rule out diffuse interstitial fibrosis or alveolitis
* History of or evidence of left-sided heart disease
* Having any other disease that is associated with pulmonary hypertension (e.g. sickle cell anemia, schistosomiasis).
* Having a musculoskeletal disorder (e.g. arthritis, artificial leg, etc.) or any other disease, which is thought to limit ambulation, or be connected to a machine, which is not portable.
* Uncontrolled systemic hypertension as evidenced by a systolic blood pressure greater than 160 millimeters of mercury (mmHg) or diastolic blood pressure greater than 100 mmHg.
* Chronic renal insufficiency as defined by serum creatinine greater than 2.5 milligrams per deciliter (mg/dL) or the requirement for dialysis.
* Receiving an investigational drug, have in place an investigational device, or have participated in an investigational drug study within the past 30 days.
* Active infection, or any other ongoing condition that would interfere with the interpretation of study assessments.
* The presence of any physiological or psychological condition that contraindicates the administration of Remodulin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Remzi Bag, MD, Principal Investigator — INTEGRIS Baptist Medical Center; Evelyn Horn, MD, Principal Investigator — Weill Medical College of Cornell University; Teresa DeMarco, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California San Francisco (UCSF) Medical Center, San Francisco, California
  - THE NEW YORK-PRESBYTERIAN HOSPITAL Weill Cornell Medical Center, New York, New York
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening was initiated by investigators at participating study sites 7 to 28 days prior to the Baseline visit. The first subject was enrolled on February 20, 2007 and the last subject completed the study on September 30, 2009. After an extended recruitment period during which no new subjects were enrolled, the study was closed in 2011.
Pre-assignment Details: A total of ten subjects were screened. Eight were enrolled and completed the study. One subject withdrew their consent prior to enrolling. The second subject failed screening due to low hemoglobin levels. Once enrolled, baseline assessments were completed, and patients underwent rapid switch from epoprostenol to treprostinil infusion.
Groups:
- Treprostinil: All Subjects transitioned from IV epoprostenol to IV treprostinil initiated to deliver a dose 20% higher than the epoprostenol dose on a ng/kg/min basis. IV treprostinil dosing was titrated without restriction during the eight week follow-up period per the investigator's judgment to optimize the dose for symptomatic benefit based on clinical signs / symptoms, exercise capacity and tolerability.
  treprostinil: rapid switch from intravenous epoprostenol on the CADD ambulatory pump to intravenous Remodulin on the Crono Five ambulatory pump
Period: Overall Study
Arm/Group | Treprostinil
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treprostinil: All Subjects transitioned from IV epoprostenol to IV treprostinil.
  treprostinil: rapid switch from intravenous epoprostenol on the CADD ambulatory pump to intravenous Remodulin on the Crono Five ambulatory pump
Arm/Group | Treprostinil
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 49.5 [45 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Pulmonary Arterial Hypertension (PAH) etiology [Number; unit: participants]
  IPAH | 6
  cardiovascular disease (CVD) | 2
Years since PAH diagnosis [Mean (Full Range); unit: years] | 7 [1.5 to 12.9]
World Health Organization (WHO) functional class at time of transition [Number; unit: participants] — WHO functional class is a system to help clinicians determine how limited a patient is in their ability to do the activities of daily living. The scale ranges from class I to class IV. In general, patients with more severe Pulmonary Hypertension (PH) tend to have a higher functional class.
  participants
    Class II | 6
    Class III | 2
epoprostenol dose [Mean (Full Range); unit: ng/kg/min] | 34.05 [7.7 to 71]
Baseline 6 Minute Walk Distance (6MWD) [Mean (Full Range); unit: meters] — This measure includes 6 patients. Two subjects did not have Baseline 6-Minute Walk Tests (6MWTs) conducted.
  meters | 390.5 [294 to 506]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 8 in 6-Minute Walk Distance (6MWD)
Description: The administration of the 6MWD test and specifications of the testing area were consistent with the American Thoracic Society guidelines and the usual practice of the investigative site [American Thoracic Society (ATS) guidelines; 2002].
Time Frame: Week 8
Population: Two subjects did not have Baseline 6MWTs and were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Treprostinil
Number analyzed (Participants) | 6
meters | -1.2 (37.0)
Statistical Analysis 1: Comparison: Treprostinil; Changes between Baseline and Week 8 were assessed using the Wilcoxon signed rank test, comparing the values at Baseline to values at Week 8. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.84, Wilcoxon signed rank

2. Secondary Outcome: Change From Baseline at Week 8 in Borg Dyspnea Score Immediately After Six Minute Walk Test
Description: The Borg dyspnea score is a 10-point scale rating the maximum level of dyspnea experienced during the 6-Minute Walk Test. Scores range from 0 (for the best condition) to 10 (for the worst condition).
Time Frame: Week 8
Population: Two subjects did not have Baseline Borg scores and were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treprostinil
Number analyzed (Participants) | 6
units on a scale | 0.08 (1.74)
Statistical Analysis 1: Comparison: Treprostinil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.00, Wilcoxon signed rank

3. Secondary Outcome: Change From Baseline at Week 8 in World Health Organization (WHO) Functional Classification
Description: WHO functional class is a system to help clinicians determine how limited a patient is in their ability to do the activities of daily living. The scale ranges from class I to class IV. In general, patients with more severe Pulmonary Hypertension (PH) tend to have a higher functional class.
Time Frame: Week 8
Population: All Subjects transitioned from IV epoprostenol to IV treprostinil were included.
Measure: Number; unit: participants
Arm/Group | Treprostinil
Number analyzed (Participants) | 8
participants
  Improved | 3
  No change | 3
  Worsened | 2
Statistical Analysis 1: Comparison: Treprostinil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.00, Wilcoxon signed rank

4. Secondary Outcome: Change From Baseline at Week 8 in Symptoms of PAH- Fatigue
Description: The presence or absence of fatigue was documented. If present, the intensity of fatigue was rated mild, moderate, or severe.
Time Frame: Week 8
Population: All Subjects transitioned from IV epoprostenol to IV treprostinil were included.
Measure: Number; unit: participants
Arm/Group | Treprostinil
Number analyzed (Participants) | 8
participants
  Improved | 1
  No change | 4
  Worsened | 3
Statistical Analysis 1: Comparison: Treprostinil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.50, Wilcoxon signed rank

5. Secondary Outcome: Change From Baseline at Week 8 in Symptoms of PAH- Dyspnea
Description: The presence or absence of dyspnea was documented. If present, the intensity of dyspnea was rated mild, moderate, or severe.
Time Frame: Week 8
Population: All Subjects transitioned from IV epoprostenol to IV treprostinil were included
Measure: Number; unit: participants
Arm/Group | Treprostinil
Number analyzed (Participants) | 8
participants
  Improved | 1
  No change | 6
  Worsened | 1
Statistical Analysis 1: Comparison: Treprostinil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.00, Wilcoxon signed rank

6. Secondary Outcome: Change From Baseline at Week 8 in Symptoms of PAH- Edema
Description: The presence or absence of edema was documented. If present, the intensity of edema was rated mild, moderate, or severe.
Time Frame: Week 8
Population: All Subjects transitioned from IV epoprostenol to IV treprostinil were included
Measure: Number; unit: participants
Arm/Group | Treprostinil
Number analyzed (Participants) | 8
participants
  Improved | 0
  No change | 6
  Worsened | 2
Statistical Analysis 1: Comparison: Treprostinil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.50, Wilcoxon signed rank

7. Secondary Outcome: Change From Baseline at Week 8 in PAH Symptoms- Orthopnea
Description: The presence or absence of orthopnea was documented. If present, the intensity of orthopnea was rated mild, moderate, or severe.
Time Frame: Week 8
Population: All Subjects transitioned from IV epoprostenol to IV treprostinil were included
Measure: Number; unit: participants
Arm/Group | Treprostinil
Number analyzed (Participants) | 8
participants
  Improved | 0
  No change | 8
  Worsened | 0
Statistical Analysis 1: Comparison: Treprostinil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.0, Wilcoxon signed rank

8. Secondary Outcome: Change From Baseline at Week 8 in PAH Symptoms- Dizziness
Description: The presence or absence of dizziness was documented. If present, the intensity of dizziness was rated mild, moderate, or severe.
Time Frame: Week 8
Population: All Subjects transitioned from IV epoprostenol to IV treprostinil were included.
Measure: Number; unit: participants
Arm/Group | Treprostinil
Number analyzed (Participants) | 8
participants
  Improved | 1
  No change | 5
  Worsened | 2
Statistical Analysis 1: Comparison: Treprostinil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.75, Wilcoxon signed rank

9. Secondary Outcome: Change From Baseline at Week 8 in PAH Symptoms- Syncope
Description: The presence or absence of syncope was documented. If present, the intensity of syncope was rated mild, moderate, or severe.
Time Frame: Week 8
Population: All Subjects transitioned from IV epoprostenol to IV treprostinil were included.
Measure: Number; unit: participants
Arm/Group | Treprostinil
Number analyzed (Participants) | 8
participants
  Improved | 0
  No change | 8
  Worsened | 0
Statistical Analysis 1: Comparison: Treprostinil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.0, Wilcoxon signed rank

10. Secondary Outcome: Change From Baseline at Week 8 in PAH Symptoms- Chest Pain
Description: The presence or absence of chest pain was documented. If present, the intensity of chest pain was rated mild, moderate, or severe.
Time Frame: Week 8
Population: All Subjects transitioned from IV epoprostenol to IV treprostinil were included.
Measure: Number; unit: participants
Arm/Group | Treprostinil
Number analyzed (Participants) | 8
participants
  Improved | 0
  No change | 7
  Worsened | 1
Statistical Analysis 1: Comparison: Treprostinil; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.00, Wilcoxon signed rank

11. Secondary Outcome: Total Weekly Time Spent With the Specific Activities Associated With Intravenous Remodulin Therapy Compared to Same Activities With Intravenous Epoprostenol
Description: A Drug Administration Activities Diary, used by subjects to record in detail the amount of time (in minutes) spent on specifically-defined drug preparation/administration activities (e.g. diluting drug, preparing reservoir, and changing tubing), was completed over a 7-day period during the Screening period while on epoprostenol and repeated at Week 7 following transition to Remodulin.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treprostinil
Number analyzed (Participants) | 8
minutes
  Gather/set-up | 4.4 (32.6)
  Prepare Drug | -50.4 (35.3)
  Connect drug | -13.1 (38.1)
  Change dressing | 3.9 (10.8)
  Total Time | -55.3 (77.0)
Statistical Analysis 1: Comparison: Treprostinil; Changes in mean times between Baseline and Week 8 were assessed using the Wilcoxon signed rank test, comparing the values at Baseline to values at Week 8. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.95, Wilcoxon signed rank — p-value for: Gather/set-up
Statistical Analysis 2: Comparison: Treprostinil; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.02, Wilcoxon signed rank — p-value for: Prepare drug
Statistical Analysis 3: Comparison: Treprostinil; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.20, Wilcoxon signed rank — p-value for: Connect drug
Statistical Analysis 4: Comparison: Treprostinil; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.48, Wilcoxon signed rank — p-value for: Change dressing
Statistical Analysis 5: Comparison: Treprostinil; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.11, Wilcoxon signed rank — p-value for: Total time

12. Secondary Outcome: Change From Baseline at Week 8 in Score on Quality of Life (QOL) Questionnaire - The Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR)
Description: The Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR), a validated PAH-specific instrument consisting of 65 items used to assess symptoms, functioning and QOL. The CAMPHOR was completed at Baseline and at Week 8. The CAMPHOR consists of 3 scales: 1. A 25-item overall symptoms scale scored 0-25, with a higher score indicating the presence of more symptoms. 2. A 15 item Activity/Functioning scale scored 0-30, where a low score indicates good functioning. 3. A 25-item QoL scale scored 0-25, with a high score indicating poor QoL. Additionally, a total score was recorded by adding up the the scores from the 3 above scales. The Symptom and QoL scales have dichotomous ('True'/'Not true') response options while the Activity/Functioning scale has three-point ('Able to do on own without difficulty'/'Able to do on own with difficulty'/'Unable to do on own') response options. The CAMPHOR score range can be from 0 to 80. A reduction in score denotes improved heath status.
Time Frame: Baseline and Week 8
Population: One subject was missing a questionnaire page of the CAMPHOR; Therefore, the component score of
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treprostinil
Number analyzed (Participants) | 8
units on a scale
  CAMPHOR- Symptom Score: number analyzed (Participants) | 7
  CAMPHOR- Symptom Score | -2.1 (4.3)
  CAMPHOR- Activity Score | 1.0 (3.9)
  CAMPHOR- Quality of Life Score: number analyzed (Participants) | 7
  CAMPHOR- Quality of Life Score | -3.1 (3.7)
  CAMPHOR- Total Score: number analyzed (Participants) | 7
  CAMPHOR- Total Score | -4.3 (10.7)
Statistical Analysis 1: Comparison: Treprostinil; Changes in mean TSQM and CAMPHOR scores between Baseline and Week 8 were assessed using the Wilcoxon signed rank test, comparing the values at Baseline to values at Week 8. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.31, Wilcoxon signed rank — p-value for: CAMPHOR Symptom Score
Statistical Analysis 2: Comparison: Treprostinil; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.84, Wilcoxon signed rank — p-value for CAMPHOR Activity Score
Statistical Analysis 3: Comparison: Treprostinil; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.03, Wilcoxon signed rank — p-value for CAMPHOR Quality of Life Score
Statistical Analysis 4: Comparison: Treprostinil; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.22, Wilcoxon signed rank — p-value for CAMPHOR Total Score

13. Secondary Outcome: Change From Baseline at Week 8 in Score on Treatment Satisfaction Questionnaire- The Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM) is a 14-question questionnaire that measures the level of satisfaction or dissatisfaction patients have with their study medication in 4 areas: effectiveness (3 questions), side effects (5 questions), convenience (3 questions), and global satisfaction (3 questions). With the exception of the first side effects question (a yes or no question), all items have 5 or 7 responses which are scored from 1 (least satisfied) to 5 or 7 (most satisfied). A total score is then summed for each domain on the following scales: effectiveness 1-21, side effects 1-20, convenience 1-21, and global satisfaction 1-17. The TSQM score range can be from 0 to 100. Lower total scores in each domain indicate dissatisfaction with the study medication and higher total scores indicate satisfaction.
Time Frame: Baseline and Week 8
Population: All 8 participants are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treprostinil
Number analyzed (Participants) | 8
units on a scale
  TSQM- Effectiveness Score | -4.9 (22.9)
  TSQM- Side-Effects Score | 7.0 (19.0)
  TSQM- Conveniences Score | 29.2 (21.4)
  TSQM- Global Satisfaction Score | -11.6 (31.7)
Statistical Analysis 1: Comparison: Treprostinil; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.55, Wilcoxon signed rank — p-value for TSQM Effectiveness Score
Statistical Analysis 2: Comparison: Treprostinil; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.50, Wilcoxon signed rank — p-value for TSQM Side-Effects Score
Statistical Analysis 3: Comparison: Treprostinil; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.01, Wilcoxon signed rank — p-value for TSQM Convenience Score
Statistical Analysis 4: Comparison: Treprostinil; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.52, Wilcoxon signed rank — p-value for TSQM Global Satisfaction Score

14. Secondary Outcome: Subject Responses to the Patient Impression of Change Questionnaire (Administered at Week 8 Only)
Description: A Patient Global Impression of Change Questionnaire, which consists of three items that ask the subject to rate changes (much better, somewhat better, about the same, somewhat worse, much worse) in their symptoms of PAH, the amount of time spent on activities associated with preparing and administering PAH therapy, and their satisfaction with their PAH therapy since transitioning from epoprostenol to intravenous Remodulin was conducted at Week 8 only and responses are reported as frequency distributions.
Time Frame: Week 8
Measure: Number; unit: participants
Arm/Group | Treprostinil
Number analyzed (Participants) | 8
participants
  Symptoms- Much Better | 4
  Symptoms- Somewhat Better | 1
  Symptoms- About The Same | 1
  Symptoms- Somewhat Worse | 1
  Symptoms- Much Worse | 1
  Time Spent- Much Less | 5
  Time Spent- Somewhat Less | 2
  Time Spent- About The Same | 0
  Time Spent- Somewhat More | 1
  Time Spent- Much More | 0
  Satisfaction- Much More Satisfied | 4
  Satisfaction- More Satisfied | 2
  Satisfaction- About The Same | 1
  Satisfaction- Less Satisfied | 0
  Satisfaction- Much Less Satisfied | 1

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were assessed upon initiation of Remodulin through to the end of study (Week 8)
Description: Since subjects were transitioning from an existing prostacyclin therapy, prostacyclin-class side effects ongoing at Baseline prior to transition were recorded separately on the specific Prostacyclin Side Effects Questionnaire. Events which increased in severity from Baseline were captured and reported as AEs.
Arm/Group | Treprostinil
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treprostinil (N=8)
central line infection (Infections and infestations) | 1 (1) — All events resolved with treatment and subjects continued in the study. The investigator judged the event to be not reasonably attributable to study drug.
Fluid overload (Cardiac disorders) | 1 (1) — One subject was hospitalized for two serious adverse events: fluid overload and right ventricular failure. All events resolved with treatment and subjects continued the study. The investigator judged the event reasonably attributable to treprostinil.
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) — All events resolved with treatment and subjects continued in the study. The investigator judged the event to be not reasonably attributable to study drug.
Right ventricular failure (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treprostinil (N=8)
Diarrhoea (Gastrointestinal disorders) | 6 (6)
Headache (Nervous system disorders) | 6 (7)
Fatigue (General disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Flushing (Vascular disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Hypotension (Vascular disorders) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Nasal congestion (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 2 (2)
Pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2)
Pyrexia (Immune system disorders) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Catheter site erythema (General disorders) | 1 (1)
Catheter site swelling (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Reproductive system and breast disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The main limitations of this study are the modest sample size and relatively short duration of follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the results of this trial must be consistent with the United Therapeutics publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.